CLINICAL TRIAL: NCT02104024
Title: Contrast Enhanced Ultrasound Scanning of Kidney and Pancreas Transplantation (Proof of Principle Study)
Brief Title: CEUS in Kidney and Pancreas Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Hussein Khambalia, Clinical research Fellow, University of Manchester
Other Study IDs: HAK 1.0
Record Dates: First submitted 2014-02-12; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Kidney Transplantation; Pancreas Transplantation
Keywords: Kidney; Pancreas; Transplant; Contrast Enhanced Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kidney transplant recipients: CEUS in Kidney Transplant recipients
  Interventions: Other: Contrast Enhanced Ultrasound Scanning
- Pancreas transplant recipients: CEUS in pancreas transplant recipients
  Interventions: Other: Contrast Enhanced Ultrasound Scanning

INTERVENTIONS:
Other: Contrast Enhanced Ultrasound Scanning
  Other Names: CEUS

SUMMARY:
This study is to investigate whether it is possible to use a special type of ultrasound scan (CEUS, Contrast Enhanced Ultrasound Scan) to view the shape, assess blood supply and calculate the amount of oxygen being carried to a transplanted kidney and pancreas. We currently use a nuclear scan (Transcan) to assess this in the kidney. This is cumbersome, involves nuclear medicine and takes 45- 60 minutes to complete.

We do not routinely image the blood supply to the pancreas post-surgery, despite the most common complication post pancreas transplantation being vascular in origin. In an emergency a CT angiogram is carried out. This involves transfer of a sick patient to the CT scanner and injection of contrast which is harmful to the kidneys.

CEUS involves injection of a safe contrast prior to conducting an ultrasound scan. This can be carried out at the bed-side, provides instant results and is cheap and safe enough to do on a routine basis for all kidney and pancreas transplant recipients. Although the uses of CEUS are well recognised, it is currently not routinely used in transplantation. CEUS has been compared to other modes of imaging and has been found to be comparable/ beneficial. However, it has never been compared to Transcan. We will therefore perform CEUS on our kidney transplant recipients and compare the results to Transcan. We will also assess whether CEUS is able to visualise the blood supply to the kidney and pancreas and quantify the perfusion to the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* adult kidney transplant recipients
* adult pancreas transplant recipients

Exclusion Criteria:

* patients unable to consent to the study
* patients under the age of 18
* patients with an absolute or relative contra-indication to receiving SonoVue contrast
* serious intra-operative complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney and pancreas transplant recipients
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
To ensure feasibility of conducting CEUS post renal and pancreas transplantation | Likely to be 24 hours post surgery.
  To ensure that conducting CEUS in the peri-operative period is logistically feasible in our centre at short-notice and it is possible to obtain images which are usable for analysis, given the presence of dressings and drains on the abdomen post surgery.
To assess patient acceptability of performing CEUS in the peri-operative period | Likely to be within 24 hours post surgery
  A validated pain questionnaire will be completed by the patient, assessing pain scores prior to and after the CEUS, compared to prior to and after the renogram.

SECONDARY OUTCOMES:
Compare the quantification (likely expressed as percentage) of organ perfusion from CEUS, with our current gold standard, the nuclear renogram. | Once both, renogram and CEUS have been performed. Likely to be within 24 hours of surgery.
  The quantification analysis of the CEUS and renograms will be correlated using descriptive statistics and either parametric or non-parametric statistical analysis to produce a correlation coefficient.
Post-operative complications | Up-to patient discharge, likely 2 weeks
  A note of all post-operative complications, up-to discharge will be assessed.

OTHER OUTCOMES:
Assess blood flow and morphology of the implanted pancreas | Likely to be within 24 hours post surgery
  Descriptive analysis of vasculature and morphology of the implanted pancreata, high-lighting potential cause of concerns eg. thrombus, bleeding, collections

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Khambalia, BMedSci, BMBS, MRCS, Principal Investigator — Manchester Royal Infirmary
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom